CLINICAL TRIAL: NCT04842500
Title: Translational Research to Inform Interventions for Severe Challenging Behavior for Individuals With Intellectual and Developmental Disabilities
Brief Title: Translational Research to Inform Interventions for Challenging Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Joseph M. Lambert, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #202204
Record Dates: First submitted 2021-04-04; First posted 2021-04-13 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: behavioral sciences; reinforcement schedule; motivation; economics, behavioral; developmental disability; intellectual disability; problem behavior; extinction bursts
MeSH Terms: conditions — Behavior; Developmental Disabilities; Intellectual Disability; Problem Behavior

STUDY DESIGN:
Intervention Model Description: The investigators will enroll 80 adults with developmental disabilities in a low-stakes translational investigation employing a 2x2 factorial, crossed, and randomized matched blocks design, with batched randomization logic. Procedures will include: (a) matching participants within batches according to progressive ratio reinforcer analysis results, and (b) randomly assigning participants to one of four experimental conditions to determine whether information about reinforcer value can be used to set baseline parameters that either promote or eliminate bursts during extinction.
Who Masked: Participant
Masking Description: Participants will be randomized to one of four baseline reinforcement conditions. They will not be informed of which condition they have been assigned to, or why they have been assigned to it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- "Cheap" Unit Price, Establishing Operation (Experimental): Pre-extinction baseline unit price for the programmed reinforcer will be its Pmax, minus one half of the distance between its Pmax and its breakpoint. Extinction will be introduced at the beginning of the relevant appointment, before within-appointment reinforcer consumption has had an opportunity to approximate demand.
  Interventions: Behavioral: Demand Informed Moderator Analysis
- "Cheap" Unit Price, Abolishing Operation (Experimental): Pre-extinction baseline unit price for the programmed reinforcer will be its Pmax, minus one half of the distance between its Pmax and its breakpoint. Extinction will be introduced at the end of the relevant appointment, after within-appointment reinforcer consumption has approximated demand.
  Interventions: Behavioral: Demand Informed Moderator Analysis
- "Expensive" Unit Price, Establishing Operation (Experimental): Pre-extinction baseline unit price for the programmed reinforcer will be its Pmax, plus one half of the distance between its Pmax and its breakpoint. Extinction will be introduced at the beginning of the relevant appointment, before within-appointment reinforcer consumption has had an opportunity to approximate demand.
  Interventions: Behavioral: Demand Informed Moderator Analysis
- "Expensive" Unit Price, Abolishing Operation (Experimental): Pre-extinction baseline unit price for the programmed reinforcer will be its Pmax, plus one half of the distance between its Pmax and its breakpoint. Extinction will be introduced at the end of the relevant appointment, after within-appointment reinforcer consumption has approximated demand.
  Interventions: Behavioral: Demand Informed Moderator Analysis

INTERVENTIONS:
Behavioral: Demand Informed Moderator Analysis — This analysis is designed to determine the degree to which relative price, and the timing of extinction, interact to increase or abate responding during extinction (thereby highlighting mechanisms of control).

SUMMARY:
This project is meant to identify relations between the reinforcement histories of 80 adults with intellectual and developmental disabilities (IDD) and the prevalence of extinction bursts. Extinction bursts, or temporary increases in rates and intensities of behavior during extinction, often preclude the inclusion of extinction in intervention packages meant to suppress severe challenging behavior, despite the fact that extinction is often necessary to generate therapeutic outcomes. Study results will provide insight into how researchers can enhance interventions for the severe challenging behavior of individuals with IDD while mitigating the undesirable collateral effects (i.e., extinction bursts) of therapeutic action (i.e., extinction). Expanded access to study results will be made available to those who inquire after all data have been obtained and analyzed.

DETAILED DESCRIPTION:
The Goal of this project is to identify mechanisms responsible for bursts, and to facilitate strategic extensions toward discovery for treatments of challenging behavior. AIM 1: In the service of this goal, the investigators aim to evaluate the accuracy of an efficient alternative to demand-curve analysis (i.e., progressive ratio reinforcer analysis) in quantifying reinforcer value (i.e., Pmax). AIM 2: Investigators also aim to evaluate the utility of manipulating baseline reinforcement parameters for controlling bursts when those manipulations are informed by the results of demand-curve analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be older than 18.
* Participants must have a developmental disability (unconstrained to specific diagnoses).
* Participants must be able to correctly manipulate all items used in the study.
* Participants must consent (or assent, when relevant) to procedures prior to and throughout the study.

Exclusion Criteria:

* Participants younger than 18.
* Participants without disabilities.
* Participants who cannot correctly manipulate items used in the study.
* Participants who do not consent (or assent, when relevant) to participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Habilitative and Training Services (HATS), Gallatin, Tennessee
  - Easterseals Tennessee: Prospect, Lebanon, Tennessee
  - Possibility Place, Murfreesboro, Tennessee
  - Next Steps at Vanderbilt, Nashville, Tennessee
  - Chrysalis, Orem, Utah

IPD SHARING:
Plan to Share IPD: Yes
Peer-reviewed published empirical reports will follow CONSORT reporting guidelines, as well as other principles of rigor and transparency highlighted through the Equator network (https://www.equator-network.org/).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, & ICF will be submitted within 12 months of study completion and will be made available indefinitely. Complete reports will be submitted for peer review within 12 months of study completion.
Access Criteria: Data and materials will be made available upon request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment entailed flyer distribution through relevant program directors. Directors vetted interest and only passed along contact information of individuals from their organization who expressed interest in the study.
Pre-assignment Details: Prior to randomization, all participants completed an assessment (i.e., the progressive-ratio analysis) that generated our matching variable (i.e., the "breakpoint" produced by the targeted reinforcer).
  Five participants dropped out during this assessment (prior to randomization). The reasons for dropping out were scheduling conflicts (x4) and a significant health concern unrelated to this study (x1).
Period: Overall Study
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
Started | 20 | 20 | 20 | 21
Completed | 15 (Note: With the exception of the implementer fidelity error, all attrition occurred prior to exposure to this study's independent variables.) | 19 (Note: With the exception of the implementer fidelity error, all attrition occurred prior to exposure to this study's independent variables.) | 18 (Note: With the exception of the implementer fidelity error, all attrition occurred prior to exposure to this study's independent variables.) | 17 (Note: With the exception of the implementer fidelity error, all attrition occurred prior to exposure to this study's independent variables.)
Not Completed | 5 | 1 | 2 | 4
Not completed — Withdrawal by Subject | 4 | 1 | 2 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation | Total
Number analyzed (Participants) | 15 | 19 | 18 | 17 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 17 | 16 | 62
  >=65 years | 2 | 3 | 1 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 5 | 6 | 29
  Male | 7 | 9 | 13 | 11 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 19 | 17 | 17 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 1 | 5
  White | 14 | 16 | 15 | 16 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 19 | 18 | 17 | 69
Disability [Count of Participants; unit: Participants] — Population: It was possible for participants to be diagnosed with more than one disability
  Participants
    Autism Spectrum Disorder | 2 | 4 | 2 | 4 | 12
    Deaf-Blindness | 0 | 0 | 0 | 0 | 0
    Deafness | 0 | 0 | 0 | 0 | 0
    Emotional Disturbance | 0 | 0 | 0 | 0 | 0
    Hearing Impairment | 0 | 0 | 0 | 0 | 0
    Intellectual Disability | 11 | 16 | 17 | 15 | 59
    Multiple Disabilities | 0 | 0 | 0 | 0 | 0
    Orthopedic Impairment | 1 | 1 | 0 | 0 | 2
    Other Health Impairment | 0 | 2 | 2 | 5 | 9
    Specific Learning Disability | 0 | 0 | 0 | 0 | 0
    Speech or Language Impairment | 0 | 1 | 1 | 0 | 2
    Traumatic Brain Injury | 2 | 0 | 0 | 0 | 2
    Visual Impairment, Including Blindness | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Peak Response Rate During Extinction
Description: This term describes the highest rate of responding observed during extinction and will be depicted as a proportion of baseline. For example, assuming the mean rate of responding during the final three sessions of baseline is 3 responses per minute (i.e., [2.8 rpm + 3.2 rpm + 3 rpm] / 3 = 3 rpm), and the highest rate of responding during a single session of extinction is 3.4 rpm, then peak response rate for this hypothetical individual would be 1.13 (i.e., 3.4 / 3 = 1.13). This value will serve as the primary dependent variable for each participant in all between-groups comparisons in our data-analysis plan.
Time Frame: This measure was obtained throughout the primary assessment (i.e., the extinction challenge)
Measure: Mean (Standard Deviation); unit: Proportion of baseline (frequency)
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
Number analyzed (Participants) | 15 | 19 | 18 | 17
Proportion of baseline (frequency) | 1.58 (1.77) | 0.85 (0.85) | 1.3 (0.87) | 0.43 (0.41)

2. Primary Outcome: Schedule Value at Breakpoint
Description: The progressive-ratio reinforcer analysis (PRA) is a game of diminishing returns that is considered an assessment of reinforcer value (e.g., if a participant does not value the reinforcer, they will quit sooner than a participant that does value the reinforcer). During the assessment, we increased the "price" (i.e., the schedule value) of reinforcers each time a participant earns two reinforcers at a currently established price.
  The breakpoint describes the "price" (schedule value; e.g., FR1, FR4, FR7) of the last obtained reinforcer prior to response cessation (i.e., the breakpoint is the last schedule value that supported enough responding to produce a reinforcer, before the participant quit playing the game). Higher breakpoints are interpreted as reflecting higher-value reinforcers. Lower breakpoints are interpreted as reflecting lower-value reinforcers.
Time Frame: PRA breakpoints were obtained during pre-assessment and were used as a matching variable prior to random assignment.
Measure: Mean (Standard Deviation); unit: Schedule Value at Breakpoint
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
Number analyzed (Participants) | 15 | 19 | 18 | 17
Schedule Value at Breakpoint | 16.45 (13.24) | 15.14 (10.21) | 16.94 (14.53) | 18.82 (15.07)

3. Primary Outcome: The Schedule Value Designated as Pmax
Description: The progressive fixed-ratio reinforcer analysis (PFRA) is an assessment of consumer demand that first establishes how much of a reinforcer a participant would consume when consumption is free of constraint (i.e., when participants can have as much of the reinforcer as they want; referred to as "bliss-point consumption").
  With bliss-point consumption established, PFRA evaluates how much a participant will "spend" (respond) to maintain bliss-point consumption patterns as price (schedule value) is increased. Unlike PRA, prices in the PFRA are held constant within each session and only increase across sessions. Initially, participants "spend" more. Eventually, they "spend" less. The price that produces maximum "spending" (i.e., higher and lower prices yield lower response outputs) is referred to as Pmax.
  Pmax is one way to quantify a reinforcer's value. That is, reinforcers that produce high Pmax have more value than reinforcers that produce low Pmax.
Time Frame: Pmax values were obtained during pre-assessment and were used as a scaling variable to set baseline schedule parameters.
Measure: Mean (Standard Deviation); unit: The Schedule Value Designated as Pmax
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
Number analyzed (Participants) | 15 | 19 | 18 | 17
The Schedule Value Designated as Pmax | 7.6 (4.42) | 7.32 (4.23) | 9 (4.12) | 7.71 (4.44)

4. Primary Outcome: Response Latency
Description: This term describes the latency from session onset to eventual response cessation during the extinction challenge.
Time Frame: This measure was obtained throughout the primary assessment (i.e., the extinction challenge)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
Number analyzed (Participants) | 15 | 19 | 18 | 17
seconds | 213.3 (185.6) | 96 (114.4) | 467.4 (607.9) | 119.8 (132.1)

5. Secondary Outcome: Number of Sessions in Extinction
Description: In addition to between-groups differences in peak-response rate (primary dependent variable), the investigators will also compare between-groups differences in the number of sessions required to achieve response elimination during extinction.
Time Frame: This measure was obtained throughout the primary assessment (i.e., the extinction challenge)
Measure: Mean (Standard Deviation); unit: Number of sessions in extinction
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
Number analyzed (Participants) | 15 | 19 | 18 | 17
Number of sessions in extinction | 1.2 (0.41) | 1.05 (0.23) | 1.89 (1.94) | 1.06 (0.24)

6. Secondary Outcome: Overall Session Duration
Description: The investigators will measure the total duration of PFRA sessions (in seconds) at Pmax to establish baseline-session parameters.
Time Frame: Duration values were obtained during pre-assessment and were used as a scaling variable to set baseline schedule parameters.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
Number analyzed (Participants) | 15 | 19 | 18 | 17
seconds | 630.87 (462.36) | 687.84 (843.27) | 668.89 (757.57) | 788.88 (930.85)

ADVERSE EVENTS:
Time Frame: Participants spent an average of 73.7 (range 5-323) calendar days completing this study. Adverse events were monitored during appointments throughout study participation.
Arm/Group | "Cheap" Unit Price, Establishing Operation | "Cheap" Unit Price, Abolishing Operation | "Expensive" Unit Price, Establishing Operation | "Expensive" Unit Price, Abolishing Operation
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/19 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/19 | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04842500/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT04842500/ICF_001.pdf